CLINICAL TRIAL: NCT01132482
Title: Phase II Study of the Effects of Sildenafil on CFTR-dependent Ion Transport Activity
Brief Title: Effects of Sildenafil on CFTR-dependent Ion Transport Activity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Jewish Health (Other)
Responsible Party: Principal Investigator, Jennifer Taylor-Cousar, Assistant Professor, National Jewish Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Sildenafil CFTR
Record Dates: First submitted 2010-04-16; First posted 2010-05-28 (Estimated); Results first posted 2019-02-26 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; CFTR; Phosphodiesterase inhibitor; Nasal potential difference; Sweat test
MeSH Terms: conditions — Cystic Fibrosis | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sildenafil (Experimental): Subjects will receive escalating doses of sildenafil
  Interventions: Drug: Sildenafil
- Placebo (Placebo Comparator): During the placebo arm, subjects receiving placebo will have sham dose escalation to maintain blinding.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil — During the course of the study, patients will receive 4 weeks of therapy: 28 days of placebo orally t.i.d. or 28 days of days of sildenafil orally t.i.d. Dosing of sildenafil will be escalated after the first week (20 mg orally t.i.d for the first week, then subjects will take 40 mg orally t.i.d. for 3 weeks). Patients not tolerating dose escalation will be discontinued from the study.
  Other Names: Revatio
  Arms: Sildenafil
Drug: Placebo — Patients receiving placebo will have sham dose escalation to maintain blinding.
  Arms: Placebo

SUMMARY:
Dehydrated airway surfaces resulting from sodium hyperabsorption and lack of chloride secretion are critical to the pathology that leads to the morbidity and mortality from Cystic Fibrosis (CF) lung disease. Previously published work in CF cell lines has demonstrated that by increasing cGMP and restoring inhibition of ENaC, sodium hyperabsorption may be reversed following administration of a phosphodiesterase inhibitor (PDEi,) such as sildenafil. Additionally it has been shown in CF cell lines and animal models, that phosphodiesterase inhibitors/analogues can enhance chloride secretion and/or correct surface localization of ΔF508 CFTR. The goal of this project is to translate the results of this work from the laboratory into a clinical trial in patients with CF using an FDA-approved therapy. The Specific Aims of this project are to: 1) Evaluate the effect of systemically administered phosphodiesterase inhibitors on ion transport in CF by measurement of Na+ and Cl- conductance by NPD and Na+ and Cl- concentration in sweat utilizing pilocarpine iontophoresis 2) To establish appropriate dosing of sildenafil in CF by performing a dose-escalation study during which patients are carefully monitored for side effects, plasma sildenafil levels are obtained and outcome measures are compared based on the dose of sildenafil administered. The results of this study in conjunction with those from an ongoing study examining the role of sildenafil as an anti-inflammatory in CF will aid in establishing safety, pharmacokinetics and mechanism of action of sildenafil in the treatment of CF lung disease.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of CF based on the following criteria: Positive sweat chloride ≥60mEq/liter (by pilocarpine iontophoresis) and genotype with two F508del CFTR mutations, and accompanied by one or more clinical features consistent with the CF phenotype
2. Male or female subjects ≥ 18 years of age
3. FEV1 ≥ 50% predicted (Hankinson)
4. Clinically stable without evidence of acute upper or lower respiratory tract infection or current pulmonary exacerbation within the 14 days prior to the screening visit
5. Ability to reproducibly perform spirometry (according to ATS criteria)
6. Ability to understand and sign a written informed consent or assent and comply with the requirements of the study
7. Willing and able to perform nasal potential difference testing
8. No changes in use of nasal medications within 2 weeks of screening visit
9. If on Orkambi, has been on stable Orkambi dose for at least 4 weeks at day 1.

Exclusion Criteria:

1. History of hypersensitivity to sildenafil
2. Use of an investigational agent within the 4-week period prior to Visit 1 (Day 0)
3. Breastfeeding, pregnant, or verbal expression of unwillingness to practice an acceptable birth control method (abstinence, hormonal or barrier methods, partner sterilization or intrauterine device) during participation in the study
4. History of significant hepatic (SGOT or SGPT > 3 times the upper limit of normal at screening, documented biliary cirrhosis, or portal hypertension), cardiovascular (history of aortic stenosis, coronary artery disease, pulmonary hypertension with right ventricular systolic pressure >55 mmHg or life-threatening arrhythmia), neurological (history of stroke), hematologic (history of bleeding diathesis), ophthalmologic (history of retinal impairment or non-arteritic ischemic optic neuritis) or renal impairment (creatinine >1.8 mg/dL.)
5. Inability to swallow pills
6. Previous lung transplantation
7. Use of concomitant nitrates, α-blocker, or Ca channel blocker
8. Use of concomitant medications known to be potent inhibitors of CYP3A4 (e.g. ketoconazole, itraconazole, ritonavir, clarithromycin, erythromycin, rifampin, verapamil)
9. Presence of a condition or abnormality that in the opinion of the investigator would compromise the safety of the subject or the quality of the data
10. Weight less than 40 kg
11. History of sputum or throat swab culture yielding Burkholderia cepacia within 2 years of screening
12. History of nasal disease or nasal surgery that would, in the opinion of the investigator, impede accurate measurements of NPD
13. Use of anticoagulant medication (e.g. heparin, coumadin)
14. Resting room air oxygen saturation <93%
15. Use of nighttime oxygen

15) History of migraine headaches 16) Baseline BP of < 90/50 mm Hg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-10; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Taylor-Cousar, MD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

REFERENCES:
- [Background] Robert R, Carlile GW, Pavel C, Liu N, Anjos SM, Liao J, Luo Y, Zhang D, Thomas DY, Hanrahan JW. Structural analog of sildenafil identified as a novel corrector of the F508del-CFTR trafficking defect. Mol Pharmacol. 2008 Feb;73(2):478-89. doi: 10.1124/mol.107.040725. Epub 2007 Nov 1. PMID 17975008
- [Background] Dormer RL, Harris CM, Clark Z, Pereira MM, Doull IJ, Norez C, Becq F, McPherson MA. Sildenafil (Viagra) corrects DeltaF508-CFTR location in nasal epithelial cells from patients with cystic fibrosis. Thorax. 2005 Jan;60(1):55-9. doi: 10.1136/thx.2003.019778. PMID 15618584
- [Background] Lubamba B, Lecourt H, Lebacq J, Lebecque P, De Jonge H, Wallemacq P, Leal T. Preclinical evidence that sildenafil and vardenafil activate chloride transport in cystic fibrosis. Am J Respir Crit Care Med. 2008 Mar 1;177(5):506-15. doi: 10.1164/rccm.200703-344OC. Epub 2007 Nov 15. PMID 18006891
- [Background] Poschet JF, Timmins GS, Taylor-Cousar JL, Ornatowski W, Fazio J, Perkett E, Wilson KR, Yu HD, de Jonge HR, Deretic V. Pharmacological modulation of cGMP levels by phosphodiesterase 5 inhibitors as a therapeutic strategy for treatment of respiratory pathology in cystic fibrosis. Am J Physiol Lung Cell Mol Physiol. 2007 Sep;293(3):L712-9. doi: 10.1152/ajplung.00314.2006. Epub 2007 Jun 22. PMID 17586695
- [Background] Poschet JF, Fazio JA, Timmins GS, Ornatowski W, Perkett E, Delgado M, Deretic V. Endosomal hyperacidification in cystic fibrosis is due to defective nitric oxide-cylic GMP signalling cascade. EMBO Rep. 2006 May;7(5):553-9. doi: 10.1038/sj.embor.7400674. Epub 2006 Apr 13. PMID 16612392
- [Background] Taylor-Cousar JL, Wiley C, Felton LA, St Clair C, Jones M, Curran-Everett D, Poch K, Nichols DP, Solomon GM, Saavedra MT, Accurso FJ, Nick JA. Pharmacokinetics and tolerability of oral sildenafil in adults with cystic fibrosis lung disease. J Cyst Fibros. 2015 Mar;14(2):228-36. doi: 10.1016/j.jcf.2014.10.006. Epub 2014 Nov 13. PMID 25466700

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sildenafil | Placebo
Started | 13 | 6
Completed | 12 | 6
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sildenafil | Placebo | Total
Number analyzed (Participants) | 12 | 6 | 18
Age, Continuous [Mean (Full Range); unit: years] | 27.1 [21 to 35] | 28 [21 to 49] | 27.6 [21 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 2 | 12
  Male | 2 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 6 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in Sodium Conductance by Nasal Potential Difference (NPD)
Description: Amount of sodium transported across the nasal epithelium
Time Frame: Baseline and day 28
Population: Patients with CF homozygous for the F508del genotype with mild, stable lung disease
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 12 | 6
mV | -0.70 (9.18) | 1.81 (7.99)

2. Secondary Outcome: Change in Chloride Conductance by NPD
Description: Amount of chloride transport across the nasal epithelium
Time Frame: Baseline and day 28
Population: Patients with CF homozygous for the F508del mutation with stable, mild lung disease
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 12 | 6
mV | 2.53 (7.58) | -0.28 (8.93)

3. Secondary Outcome: Change in Sweat Chloride Concentration by Pilocarpine Iontophoresis
Description: Amount of chloride transport across the skin
Time Frame: Baseline and day 28
Population: Patients with CF homozygous for the F508del mutation with mild, stable lung disease. One patient in the sildenafil group had insufficient sweat for analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 11 | 6
mmol/L | 6.13 (14.4) | -0.42 (11.91)

4. Secondary Outcome: Change in Pulmonary Function by Spirometry
Description: ppFEV1
Time Frame: Baseline and day 28
Population: Patients with CF homozygous for the F508del mutation with mild, stable lung disease
Measure: Mean (Standard Deviation); unit: % predicted
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 12 | 6
% predicted | -0.92 (6.53) | -1.00 (3.69)

5. Secondary Outcome: Change in Serum Sildenafil Pharmacokinetics
Description: Trough sildenafil levels
Time Frame: Baseline and day 28
Population: Patients with CF homozygous for the F508del mutation with mild, stable lung disease
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 12 | 6
ug/mL | 0 (0) | 0 (0)

6. Secondary Outcome: Change in CF Heath Related Quality of Life Questionnaire (CFQ-R)
Description: Respiratory domain of the CFQ-R; The range of scores is 0-100, with higher scores indicating better health.
Time Frame: Baseline and day 28
Population: Patients with CF homozygous for the F508del mutation with mild, stable lung disease
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 12 | 6
units on a scale | -1.87 (14.26) | 0.00 (14.04)

7. Secondary Outcome: Change in Lung Clearance Index
Description: The lung clearance index (LCI) measures how long it takes for an inert gas (e.g. nitrogen) to be washed out of the lungs during relaxed tidal breathing. A higher value of the LCI indicates worse disease. LCI is calculated as the number of functional residual capacity (FRC) turnovers required to reduce the end-tidal concentration of nitrogen to 1/40th of the starting concentration and is calculated by dividing the sum of exhaled tidal breaths (cumulative exhaled volume (CEV)) by simultaneously measured FRC.
Time Frame: Baseline and day 28
Population: Patients with CF homozygous for the F508del mutation with mild, stable lung disease who had valid data for measure
Measure: Mean (Standard Deviation); unit: LCI
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 9 | 5
LCI | -0.33 (1.77) | -1.14 (2.94)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of screening to 1 week following the last dose of study drug (approximately 2 months).
Arm/Group | Sildenafil | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/6
Other Adverse Events (participants affected / at risk) | 10/12 | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sildenafil (N=12) | Placebo (N=6)
DIOS (Gastrointestinal disorders) | 1 (1) | 0 (0) — Distal Intestinal Obstruction Syndrome
Pulmonary exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sildenafil (N=12) | Placebo (N=6)
Pain, throat (General disorders) | 2 (2) | 0 (0) — Sore throat
Pain, head (General disorders) | 5 (7) | 0 (0) — Headache
Rhinorrhea (General disorders) | 2 (2) | 1 (1) — Runny nose/sinus drainage
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) — myalgia, achiness
Flushing (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pain, chest (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) — Chest heaviness with exertion
Heartburn (Gastrointestinal disorders) | 1 (1) | 1 (1) — Dyspepsia
cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Elevated ALT (Gastrointestinal disorders) | 1 (1) | 0 (0)
Elevated AST (Gastrointestinal disorders) | 1 (1) | 0 (0)
Distension/bloating, abdominal (Gastrointestinal disorders) | 0 (0) | 1 (1) — Distention
upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — URI
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Pulmonary exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Increased sputum clearance (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was a small, single center one. However, the study was appropriately powered to detect a differences in the primary outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-21): https://cdn.clinicaltrials.gov/large-docs/82/NCT01132482/Prot_SAP_000.pdf